CLINICAL TRIAL: NCT04297254
Title: A Prospective, Multicenter, Post-marketing Phase IV Study to Assess the Safety and Efficacy of Lenvatinib as First-line Treatment in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: A Study to Assess the Safety and Efficacy of Lenvatinib as First-line Treatment in Participants With Unresectable HCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Pharmaceuticals India Pvt. Ltd (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-M091-511
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Lenvatinib; E7080; Unresectable hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib 12 mg or 8 mg (Experimental): Participants with body weight (BW) greater than or equal to (>=) 60 kilogram (kg), will receive lenvatinib 12 milligram (mg) (03 capsules), and participants with BW less than (<) 60 kg, will receive lenvatinib 8 mg, (02 capsules), orally, once daily with or without food in 28-day cycles for a maximum 6 cycles of 4 weeks each for a total of 24 weeks or until disease progression, death, intolerable or unacceptable toxicity, or withdrawal of consent, whichever occurs earlier.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsules.

SUMMARY:
The primary objective of this study is to evaluate the safety of lenvatinib in HCC.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, single-arm, non-comparative, post-marketing phase IV study. This study will enroll 50 participants with unresectable HCC. Participants will receive lenvatinib for 24 weeks or until disease progression, death, intolerable or unacceptable toxicity, or withdrawal of consent, whichever occurs earlier. All participants will be followed up for an end-of-study (EOS) visit at 4 weeks after the completion of 24 weeks of treatment or after last treatment visit if earlier, as applicable that is end-of-treatment (EOT).

Participants who completed 24 weeks of therapy and continue to show clinical benefit will be able to continue to receive lenvatinib (beyond week 24 as necessary) as per Investigator's discretion and based on radiological response.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of >=18 years of age
2. Participant or their legally acceptable representative (LAR) is willing to sign written informed consent for participation in the study and ready to comply with the study procedures and schedule
3. Must have a confirmed diagnosis of unresectable HCC with one of the following criteria:

   * Histologically or cytologically confirmed diagnosis of HCC
   * Clinically confirmed diagnosis of HCC according to the American Association for the Study of Liver Diseases (AASLD) criteria, including cirrhosis of any aetiology or with chronic hepatitis B or C infection criteria
4. At least 1 measurable target lesion according to RECIST 1.1 meeting the following criteria:

   * Hepatic lesion:

     * The lesion can be accurately measured in at least one dimension as >=1.0 centimeter (cm)
     * The lesion is suitable for repeat measurement
   * Non-hepatic lesion:

     * Lymph node (LN) lesion that measures at least one dimension as >=1.5 cm in the short axis, except for porta hepatis LN that measures >=2.0 cm in the short axis
     * Non-nodal lesion that measures >=1.0 cm in the longest diameter
   * Lesions previously treated with radiotherapy or locoregional therapy must show radiographic evidence of disease progression to be deemed a target lesion
5. Participants are categorized to Stage B (not applicable for transarterial chemoembolization [TACE]) or Stage C based on Barcelona Clinic Liver Cancer (BCLC) staging system.
6. Has adequate bone marrow function, defined as:

   * Absolute neutrophil count (ANC) >= 1.5*10^9 per liter (/L)
   * Haemoglobin >=8.5 gram per deciliter (g/dL)
   * Platelet count >=75*10^9/L
7. Adequate liver function based on liver function tests, defined as:

   * Albumin >=2.8 g/dL
   * Bilirubin less than or equal to <=3.0 milligram per deciliter (mg/dL)
   * Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine aminotransferase (ALT) <=5*the upper limit of normal (ULN)
8. Adequate blood coagulation function, defined as international normalized ratio (INR) <=2.3
9. Adequate renal function, defined as >30 milliliter per minute (ml/min) calculated as per the Cockcroft and Gault formula
10. Adequately controlled blood pressure (BP) with 0 or 1 antihypertensive medications, defined as BP <=150/90 millimeter of mercury (mmHg) at screening and no change in antihypertensive medications within 1 week before Cycle 1 Day 1
11. Adequate pancreatic function, defined as amylase and lipase <=1.5*ULN
12. With a Child-Pugh score A
13. With Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
14. With life expectancy of >=12 weeks from the start of study treatment, as per Investigator's judgement.

Exclusion Criteria:

1. With imaging findings for HCC corresponding to any of the following:

   * HCC with >=50% liver occupation
   * Clear invasion into the bile duct
   * Portal vein invasion at the main portal branch (Vp4)
2. Who have received any systemic chemotherapy, including sorafenib, or immunotherapy, or any systemic investigational anticancer agents for advanced/unresectable HCC
3. Who have received any anticancer therapy (including surgery, percutaneous ethanol injection, radio frequency ablation, transarterial [chemo] embolization, hepatic intra-arterial chemotherapy, biological, immunotherapy, hormonal, or radiotherapy) or any blood enhancing treatment (including blood transfusion, blood products, or agents that stimulate blood cell production, example granulocyte colony-stimulating factor [G-CSF]) within 28 days prior to enrolment
4. Who have not recovered from toxicities as a result of prior anticancer therapy, except alopecia and infertility
5. With significant cardiovascular impairment including but not limited to the history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within previous 6 months, or cardiac arrhythmia requiring medical treatment at the time of screening
6. With prolongation of corrected QT (QTc) interval to >480 millisecond (ms)
7. With gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib in the opinion of the Investigator
8. Bleeding or thrombotic disorders or use of anticoagulants such as, warfarin or similar agents requiring therapeutic international normalized ratio (INR) monitoring
9. Having a gastrointestinal bleeding event or active haemoptysis (bright red blood of at least 0.5 teaspoon) within 28 days prior to enrollment
10. With gastric or oesophageal varices that may require treatment
11. With any other active malignancy (except for HCC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 36 months prior to enrolment
12. Any history of, or concurrent, brain or subdural metastases
13. Having >1 + proteinuria on urine dipstick testing will undergo 24 hour (h) urine collection for quantitative assessment of proteinuria. Patients with urine protein >=1 gram per 24 hour (g/24 h) will be excluded
14. With arterial-portal venous shunt or arterial-venous shunt preventing a proper diagnosis of the tumour
15. Any medical or other condition that in the opinion of the Investigator would preclude the participant's participation in the study.
16. With known intolerance to lenvatinib (or any of the excipients)
17. With positive human immunodeficiency virus (HIV) or active infection requiring treatment (except for hepatitis virus)
18. Who cannot be evaluated by either triphasic liver computed tomography (CT) or triphasic liver magnetic resonance imaging (MRI) because of allergy or other contraindication to both CT and MRI contrast agents
19. Have undergone major surgery within 3 weeks prior to the entry in the study or are scheduled for a surgery during the study period
20. Have already undergone a liver transplant
21. Female participants who are breastfeeding or pregnant at the time of enrolment in the study
22. Female participants of childbearing potential who, within 4 weeks prior to study enrolment, did not use a highly effective method of contraception or do not agree to use a highly effective method of contraception throughout the study period
23. Current abuse of alcohol; and current or past (last 12 months) abuse of drugs
24. Participation in a concurrent clinical trial or in another trial within the 6 months prior to this study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Grade 3 or Higher Treatment-emergent Adverse Events (TEAEs) | Baseline up to Week 24
  TEAEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. The severity of all adverse events (AEs) will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The grades are: Grade 1 (Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily life [ADL]); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 (Life-threatening consequences; urgent intervention indicated); and Grade 5 (Death related to AE).
Number of Participants with Serious Adverse Events (SAEs) | Baseline up to Week 24
Number of Participants with Grades 1 and 2 Treatment-emergent Adverse Events (TEAEs) | Baseline up to Week 24
  TEAEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. The severity of all AEs will be graded according to CTCAE version 4.0. The grades are: Grade 1 (Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 (Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL); Grade 3 (Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 (Life-threatening consequences; urgent intervention indicated); and Grade 5 (Death related to AE).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From the start of study treatment up to Week 24
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as the best overall response from the start of study treatment up to Week 24. CR per response evaluation criteria in solid tumor (RECIST) 1.1 is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR per RECIST 1.1 is defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Progression-free Survival (PFS) | From date of first dose of study drug until documentation of disease progression or death from any cause (whichever occurs first) or up to approximately Week 24
  PFS is defined as the time from the start of treatment until the first occurrence of disease progression (PD) or death, whichever is earlier. PD per RECIST 1.1 is defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Percentage of Participants Requiring Dose Modifications (Dose Interruptions or Dose Reductions) | Baseline up to Week 24
Time to First Dose Reduction | Baseline up to Week 24

CONTACTS AND LOCATIONS:
Locations (10):
- India (10):
  - HCG Comprehensive Cancer Care Hospital, Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Shatabdi Hospital, Nashik, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - LMMF's Deenanath Mangeshkar Hospital & Research Center, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Somani Hospital, Jaipur, Rajasthan
  - Meenakshi Mission Hospital, Madurai, Tamil Nadu
  - Apollo Gleneagles Hospital Limited, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.